CLINICAL TRIAL: NCT03916731
Title: First in Human Evaluation of STARgraft AV for Hemodialysis Access in Comparison to ePTFE Vascular Grafts
Brief Title: Evaluation of STARgraft AV for Hemodialysis Access
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Healionics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIP 00355
Record Dates: First submitted 2019-04-08; First posted 2019-04-16 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: End Stage Renal Disease
Keywords: Hemodialysis; Vascular Access; Arterio-Venous Grafts (AVG)
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: Equal numbers of Participants are randomly assigned investigational or control grafts for implant. Study follow up examinations and routine dialysis procedures over the study period are identical for both groups.
Who Masked: Participant, Care Provider
Masking Description: Randomized Assignment of Investigational and Control devices by Sponsor. Participants and Dialysis Clinics providing routine maintenance hemodialysis care are masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- STARgraft AV (Experimental): Participants will be implanted with 6mm diameter STARgraft AV grafts as an upper arm Brachial Artery to Axillary Vein shunt for hemodialysis access.
  Interventions: Device: STARgraft AV
- Control (ePTFE) (Active Comparator): Participants will be implanted in the same upper arm location with standard 6mm diameter ePTFE dialysis access grafts. All other aspects of this study arm are identical to the Experimental one.
  Interventions: Device: ePTFE AV graft (control)

INTERVENTIONS:
Device: STARgraft AV — Implant of STARgraft AV shunt in the upper arm and subsequent use for hemodialysis access. After healing from the surgical procedure the graft will be routinely cannulated for hemodialysis sessions. Periodic evaluations of blood flow by ultrasound imaging will be made over the study period. Established standards of care will be followed as needed to maintain dialysis function.
  Arms: STARgraft AV
Device: ePTFE AV graft (control) — Implant of standard ePTFE AV shunt as a control in the upper arm and subsequent use for hemodialysis access. After healing from the surgical procedure the graft will be routinely cannulated for hemodialysis sessions. Periodic evaluations of blood flow by ultrasound imaging will be made over the study period. Established standards of care will be followed as needed to maintain dialysis function.
  Arms: Control (ePTFE)

SUMMARY:
This study is a First-in-Human, single site, prospective, randomized, controlled evaluation of the safety and effectiveness of the Healionics STARgraft AV hemodialysis access graft. The STARgraft has been demonstrated in preclinical studies to have improved resistance to the common failure mode of venous anastomosis stenosis.

Performance of the STARgraft AV will be compared against control implants of commercially available standard ePTFE grafts approved for the same use.

The study is enrolling patients with End Stage Renal Disease (ESRD) requiring hemodialysis via a prosthetic vascular graft. The study proposes to:

1. Demonstrate improved primary patency of the investigational STARgraft AV compared to the ePTFE controls over a period of 6 months, with extended results to 1 year.
2. Verify safety of the STARgraft AV multilayer construction in extended vascular access use.

It is intended to enroll 25 subjects each for the investigational devices and the controls respectively (50 total) with randomized device allocation at subject presentation for implant surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, > 18 years or age.
2. Patient has given informed consent to participate in the trial.
3. Stated willingness to comply with all study procedures and availability for the duration of the study.
4. Able to effectively communicate with study personnel.
5. Candidate for a new arterio-venous graft placed in the upper arm.
6. Life expectancy judged to be at least 2 years.
7. Axillary vein of greater than or equal to 7 mm in diameter.
8. Brachial artery of greater than or equal to 4 mm in diameter.
9. Systolic blood pressure equal to or greater than 120 mmHg.
10. Absence of central venous stenosis downstream from implant site confirmed with ultrasound and/or angiogram.

Exclusion Criteria:

1. Unable or unlikely to comply with trial protocol and/or follow-up.
2. Pregnancy.
3. Clinical morbid obesity.
4. Anatomical limitations.
5. Immunodeficiency syndrome.
6. History of bacterial infection within 8 weeks prior to graft implantation.
7. History of hypercoagulation or bleeding disorders.
8. Elevated platelet count > 1 million per microliter of blood.
9. History of heparin-induced thrombocytopenia syndrome (HIT).
10. Medically confirmed stenosis of the veins downstream of the implant site.
11. Inadequate arterial flow or pressure proximal to the implant site.
12. Currently participating in another investigation drug or device study which may clinically interfere with any endpoints of this trial.
13. Fever greater than 38° C.
14. Prior allergic reaction to silicone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2020-10-17 (Actual); Study Completion 2021-05-11 (Actual)

PRIMARY OUTCOMES:
Primary Unassisted Patency | 12 months post implantation.
  Percentage of subjects without an occurrence of either an access thrombosis or an access procedure performed to maintain patency.

SECONDARY OUTCOMES:
Primary Unassisted Patency | 1, 2, 4, 9 and 12 months post implantation
  Percentage of subjects without an occurrence of either an access thrombosis or an access procedure performed to maintain patency.
Assisted Primary Patency | 1, 2, 4, 6, 9 and 12 months post implantation
  Percentage of subjects retaining patency after one or more interventions so long as patency was not lost at any point.
Secondary Patency (Cumulative Patency) | 1, 2, 4, 6, 9 and 12 months post implantation
  Percentage of subjects without loss of access at the original implant site.
Graft Related Infections | 1, 2, 4, 6, 9 and 12 months post implantation
  Frequency of infections related to graft placement and use for dialysis access.
Safety Outcomes | 1, 2, 4, 6, 9 and 12 months post implantation
  Frequency and Severity of Adverse Events resulting from graft implantation and use for hemodialysis access.

OTHER OUTCOMES:
Blood flow rates in grafts. | 2 weeks and 1, 2, 4, 6, 9, 12 months post implantation.
  Ultrasound measurements of flow rates (ml/minute) to detect patency trends with time after implantation
Peak Systolic Velocity (PSV) Ratio | 2 weeks and 1, 2, 4, 6, 9, 12 months post implantation
  Ultrasound measurement of PSV (The ratio of flow velocity at the venous anastomosis to that at a point 2cm upstream in the graft)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Ebner, MD, Principal Investigator — Italian Hospital Asuncion Paraguay
Locations (1):
- Italian Hospital, Asunción, Paraguay

IPD SHARING:
Plan to Share IPD: No